CLINICAL TRIAL: NCT04441606
Title: The Role of 68Ga-FAPI-04 PET/CT as a Problem Solving Imaging Modality in Various Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-20-ES-0308-CTIL
Record Dates: First submitted 2020-06-14; First posted 2020-06-22 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2020-06

CONDITIONS: Different Types of Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Different types of cancer (Experimental): The study population will include up to 50 patients with disease in whom a diagnostic challenge is met, including but not limited to:
  1. Inconclusive findings on 18F-FDG PET/CT or other imaging modalities.
  2. Better delineation of tumor extent prior to therapy
  3. Malignancies known to show variable avidity to FDG and at times, no uptake at all (e.g. Exocrine Pancreatic cancer, Gastric carcinoma, Mucin-producing or Signet-ring carcinoma).
  4. Patients unable to optimally comply with the required preparation for FDG imaging.
     * The study population will include only patients treated in Tel-Aviv Sourasky Medical Center, Tel-Aviv, Israel, and referred by their attending physicians, of whom are part of the hospital staff.
  Interventions: Radiation: 68Ga-FAPI-04 PET/CT

INTERVENTIONS:
Radiation: 68Ga-FAPI-04 PET/CT — * Patients will undergo two scans: first a routine FDG PET scan and a FAPI PET scan, within 10 days.
  * Scans will be interpreted by board certified Nuclear medicine physicians and board certified radiologists.
  * Immunohistochemical analysis with specific staining for FAP will be performed in removed malignant tissues, either at surgery or from biopsy, to assess a possible correlation between the intensity of uptake and the level of FAP expression.

SUMMARY:
The aim of the suggested study is to assess the added value of 68Ga-FAPI-04 PET/CT over 18F-FDG PET/CT in evaluating the extent of disease in patients with various malignancies, in whom a diagnostic challenge is met, such as inconclusive findings on 18F-FDG PET/CT or other imaging studies, better delineation of tumor extent prior to therapy, and with emphasis on malignancies known to show variable avidity to FDG and at times, no uptake at all. Also patients unable to optimally comply with the required preparation for FDG imaging, such as diabetic patients who struggle in achieving glycemic control.

ELIGIBILITY:
Inclusion Criteria:

The study population will include up to 50 patients with disease in whom a diagnostic challenge is met, including but not limited to:

1. Inconclusive findings on 18F-FDG PET/CT or other imaging modalities.
2. Better delineation of tumor extent prior to therapy
3. Malignancies known to show variable avidity to FDG and at times, no uptake at all (e.g. Exocrine Pancreatic cancer, Gastric carcinoma, Mucin-producing or Signet-ring carcinoma).
4. Patients unable to optimally comply with the required preparation for FDG imaging.

   * The study population will include only patients treated in Tel-Aviv Sourasky Medical Center, Tel-Aviv, Israel, and referred by their attending physicians, of whom are part of the hospital staff.

Exclusion Criteria:

* Age < 18 years.
* Pregnant females.
* Patients who are reluctant to undergo both FDG and FAPI PET scans.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Patients who preformed 68Ga-FAPI-04 PSMA. | 1 year
  To evaluate the avidity of various cancers to 68Ga-FAPI-04.
Patients who preformed 68Ga-FAPI-04 PSMA and PET/CT FDG. | 1 year
  To compare the detectability of FAPI-04 and FDG for malignant lesions.
Patients who preformed 68Ga-FAPI-04 PSMA and PET/MRI. | 1 year
  To evaluate the potential impact of 68Ga-FAPI-04 PET/CT and/or PET/MRI on patient management.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky medial center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided